CLINICAL TRIAL: NCT00666848
Title: Effect of Sitagliptin on the Blood Pressure Response to ACE Inhibition in the Metabolic Syndrome
Brief Title: Effect of Sitagliptin and an ACE Inhibitor on Blood Pressure in Metabolic Syndrome
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Vanderbilt University (Other)
Responsible Party: Principal Investigator, Nancy J. Brown, Robert H. Williams Professor of Medicine and Pharmacology, Vanderbilt University
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: 070977
Record Dates: First submitted 2008-04-23; First posted 2008-04-25 (Estimated); Results first posted 2012-05-11 (Estimated); Last update posted 2012-05-11 (Estimated); Status verified 2012-04

CONDITIONS: Metabolic Syndrome; Hypertension
Keywords: Metabolic syndrome; Hypertension; Sitagliptin; Enalapril
MeSH Terms: conditions — Metabolic Syndrome; Hypertension | interventions — Enalapril; Sitagliptin Phosphate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- 2 (enalapril 5mg) (Placebo Comparator): Subjects received Enalapril 5mg on study day and a placebo pill for 5 days prior or subjects received enalapril 5mg on study day and sitagliptin 100mg/day for 5 days prior .
  Interventions: Drug: Enalapril 5mg; Drug: Sitagliptin
- 1 (placebo) (Placebo Comparator): Subjects received a placebo pill on study day and received a placebo pill for 5 days prior or subjects received a Placebo pill on study day and sitagliptin 100mg for 5 days prior.
  Interventions: Drug: Placebo; Drug: Sitagliptin
- 3 (enalapril 10mg) (Placebo Comparator): Subjects received Enalapril 10mg on study day and a placebo pill for 5 days prior, or subjects received Enalapril 10mg on study day and sitagliptin 100mg for 5 days prior.
  Interventions: Drug: Enalapril 10mg; Drug: Sitagliptin

INTERVENTIONS:
Drug: Placebo — Enalapril 0mg after 5 days of placebo versus after 5 days sitagliptin 100mg/d
  Arms: 1 (placebo)
Drug: Enalapril 5mg — Enalapril 5 mg after 5 days placebo versus after 5 days sitagliptin 100mg/d
  Arms: 2 (enalapril 5mg)
Drug: Enalapril 10mg — Enalapril 10mg after 5 days placebo versus after 5 days sitagliptin 100 mg/d
  Arms: 3 (enalapril 10mg)
Drug: Sitagliptin — Sitagliptin 100mg/day for 5 days crossed over to placebo daily for 5 days prior to arms.

SUMMARY:
This study will measure the effect of the anti-diabetic agent sitagliptin on blood pressure in individuals with the metabolic syndrome. We will also measure the effect of sitagliptin on blood pressure in people already taking a blood pressure medication called an ACE inhibitor.

DETAILED DESCRIPTION:
The prevalence of metabolic syndrome and Type 2 diabetes mellitus (T2DM) has reached epidemic proportions in developed countries and is closely associated with hypertension. As new oral hypoglycemic agents become available for clinical use, practitioners wishing to treat both hyperglycemia and hypertension will use varieties of combinations of medications. In this setting, understanding interactions and additive effects of these medications becomes essential. Sitagliptin, a selective dipeptidyl peptidase-IV (DPP-4) inhibitor, improves glycemic control in patients with T2DM by decreasing the degradation of the incretin hormones. The incretin hormones glucagon-like peptide-1 (GLP-1) and glucose-dependent insulinotropic peptide (GIP) augment nutrient mediated insulin release. To date there have been two reports of a blood pressure lowering effect of the DPP-4 inhibitor vildagliptin, but no mechanism for this effect has been proposed.

Specific Aim 1: To test the hypothesis that the DPP-4 inhibitor sitagliptin lowers blood pressure compared to placebo therapy in subjects with the metabolic syndrome.

Specific Aim 2: To test the hypothesis that the DPP-4 inhibitor sitagliptin potentiates the blood pressure response to acute ACE-inhibition.

ELIGIBILITY:
Inclusion Criteria:

* Ambulatory subjects, 18 to 70 years of age, inclusive
* For female subjects, the following criteria must be met:

  * Postmenopausal for at least 1 year, or
  * Status-post surgical sterilization, or
  * If of childbearing potential, utilization of barrier contraceptive and willingness to undergo beta-hcg testing prior to drug treatment and on every study day
* Metabolic syndrome as defined by 3 or more of the following:

  * Fasting plasma glucose of at least 100 mg/dL (5.6 mmol/L)
  * Serum triglycerides of at least 150 mg/dL (1.7 mmol/L)
  * Serum HDL less than or equal to 40 mg/dL in men or less than 50 mg/dL in women or on cholesterol-lowering medications
  * Blood pressure of at least 130/85 mmHg or on blood-pressure lowering medications
  * Waist girth of more than 102 cm in med or 88 cm in women
* Statin therapy for hypercholesterolemia must be a steady dose for 6 months prior to study day

Exclusion Criteria:

* Diabetes type 1 or type 2, as defined by a fasting glucose of 126 mg/dL or greater or the use of anti-diabetic medication
* History of reported or recorded hypoglycemia (plasma glucose less than 70 mg/dL)
* Use of hormone replacement therapy
* In hypertensive patients, a seated systolic blood pressure greater than 179 mmHg or a seated diastolic blood pressure greater than 110 mmHg
* Pregnancy
* Breast-feeding
* Cardiovascular disease such as myocardial infarction within 6 months prior to enrollment, presence of angina pectoris, significant arrhythmia, congestive heart failure (LV hypertrophy acceptable), deep vein thrombosis, pulmonary embolism, second or third degree heart block, mitral valve stenosis, aortic stenosis or hypertrophic cardiomyopathy
* Treatment with anticoagulants
* History of serious neurological disease such as cerebral hemorrhage, stroke, or transient ischemic attack
* History or presence of immunological or hematological disorders
* Diagnosis of current asthma
* History of angioedema associated with use of ACE-I
* Clinically significant gastrointestinal impairment that could interfere with drug absorption
* Impaired hepatic function (aspartate amino transaminase [AST] and/or alanine amino transferase [ALT] > 2.0 x upper limit of normal range)
* Impaired renal function (serum creatinine > 1.5 mg/dl)
* Hematocrit <35%
* Any underlying or acute disease requiring regular medication which could possibly pose a threat to the subject or make implementation of the protocol or interpretation of the study results difficult
* Treatment with chronic systemic glucocorticoid therapy (more than 7 consecutive days in 1 month)
* Treatment with lithium salts
* History of alcohol or drug abuse
* Treatment with any investigational drug in the 1 month preceding the study
* Mental conditions rendering the subject unable to understand the nature, scope and possible consequences of the study
* Inability to comply with the protocol, e.g. uncooperative attitude, inability to return for follow-up visits, and unlikelihood of completing the study
* Oral contraceptives

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2008-03; Primary Completion 2009-08 (Actual); Study Completion 2010-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Nancy J Brown, M.D., Principal Investigator — Vanderbilt University Medical Center
Locations (1):
- Vanderbilt University Medical Center, Nashville, Tennessee, United States

REFERENCES:
- [Result] Marney A, Kunchakarra S, Byrne L, Brown NJ. Interactive hemodynamic effects of dipeptidyl peptidase-IV inhibition and angiotensin-converting enzyme inhibition in humans. Hypertension. 2010 Oct;56(4):728-33. doi: 10.1161/HYPERTENSIONAHA.110.156554. Epub 2010 Aug 2. PMID 20679179

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Subjects received a placebo pill for 5 days prior then arm 1,2,or3 and crossed over to sitagliptin 100mg/day for 5 days prior to arm 1,2,or3. This is a parallel cross over study. 43 subjects were consented. 15 did not meet inclusion criteria. 3 withdrew before randomization.
Period: Overall Study
Arm/Group | 2 (Enalapril 5mg) | 1 (Placebo) | 3 (Enalapril 10mg)
Started | 8 (15 didn't meet inclusion criteria. 3 withdrew before randomized. 1 withdrawn before randomized.) | 9 (15 didn't meet inclusion criteria. 3 withdrew before randomized. 1 withdrawn before randomized.) | 7 (15 didn't meet inclusion criteria. 3 withdrew before randomized. 1 withdrawn before randomized.)
Completed | 8 (finished Aim 2) | 9 (finished Aim 1) | 7 (finished Aim 3)
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | 2 (Enalapril 5mg) | 1 (Placebo) | 3 (Enalapril 10mg) | Total
Number analyzed (Participants) | 8 | 9 | 7 | 24
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 8 | 8 | 7 | 23
  >=65 years | 0 | 1 | 0 | 1
Age Continuous [Mean (Standard Deviation); unit: years] | 42 (9.8) | 44 (13.9) | 41 (9.1) | 43 (2.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 4 | 4 | 11
  Male | 5 | 5 | 3 | 13
Region of Enrollment [Number; unit: participants]
  United States | 8 | 9 | 7 | 24

OUTCOME MEASURES:

1. Primary Outcome: Change in MAP During Placebo
Description: The change in mean arterial pressure (MAP) in response to placebo or enalapril after pretreatment with 5 days of placebo
Time Frame: just prior to drug administration and 8 hours after drug administration
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | 2 (Enalapril 5mg) | 1 (Placebo) | 3 (Enalapril 10mg)
Number analyzed (Participants) | 8 | 9 | 7
mmHg | -0.9 (2.5) | 2.7 (2.1) | -7.9 (2.4)

2. Primary Outcome: Change in MAP During Sitagliptin
Description: Mean change in mean arterial pressure in response to placebo or enalapril in the presence of 5 days of sitagliptin 100mg/day
Time Frame: just prior to drug administration and 8 hours following treatment
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | 2 (Enalapril 5mg) | 1 (Placebo) | 3 (Enalapril 10mg)
Number analyzed (Participants) | 8 | 9 | 7
mmHg | -5.7 (2.0) | -2.3 (2.0) | -0.9 (2.3)

ADVERSE EVENTS:
Time Frame: 2 years.
Arm/Group | 2 (Enalapril 5mg) | 1 (Placebo) | 3 (Enalapril 10mg)
Serious Adverse Events (participants affected / at risk) | 0/8 | 0/9 | 0/7
Other Adverse Events (participants affected / at risk) | 0/8 | 0/9 | 0/7

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No